CLINICAL TRIAL: NCT05275712
Title: Outcome of Cochlear Implant in Children at Assiut University Hospital
Brief Title: Outcome of Cochlear Implant in Assiut University
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Sally Shenouda Bolis, Resident doctor, Assiut University
Other Study IDs: Outcome of cochlear implant
Record Dates: First submitted 2022-03-01; First posted 2022-03-11 (Actual); Last update posted 2023-02-22 (Actual); Status verified 2022-03

CONDITIONS: Cochlear Implant

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Audiological evaluation — Questionnaire for parents about their children behavior after implantation, audiological evaluation and speech perception test .

SUMMARY:
Evaluation of the outcome of cochlear implanted children at audiovestibular medicine unit in Assiut university hospital.

DETAILED DESCRIPTION:
Hearing loss is one of the most common health problems affecting people around the world with an average international incidence of 5% .

In Egypt, it affects 16% of the population with an incidence of 14% in children less than 14 years old. 86% of deaf patients had conductive hearing loss (CHL), while sensorineural hearing loss (SNHL) was found in 14%, with a male to female ratio of 3:2 HL .

Cochlear implantation (CI) has become a routine procedure in the United States and worldwide for the management of severe-to-profound SNHL loss. It is a remarkable example of success that was made possible through collaboration between engineers, surgeons, scientists and the medical community .

Early cochlear implantation had a long-term positive impact on auditory and verbal development, if auditory stimulation does not occur within this timeframe, the auditory system degenerates. It has been suggested that in the absence of normal auditory stimulation there is a period of about 3.5 years during which the central auditory system retains its maximum plasticity. This can extend in some children up to the age of approximately 7 years, after which it is significantly reduced. The earlier implantation causes better outcomes, including improved language development, speech perception and speech production skills .

Early research reviews found that the ability to communicate in spoken language was better the earlier the implantation was performed. These reviews also found that cochlear implants provide open set speech understanding for the majority of implanted profoundly hearing-impaired children, and that it was not possible to accurately predict the specific outcome of the given implanted child .

Research since then has reported long-term socio-economic benefits for children as well as audiological outcomes including improved sound localization and speech perception .

The outcome of CI surgery on Quality of Life (QoL) has been greatly investigated via parental questionnaire assessment. This questionnaire was designed with 11 subscales and 58 questions in total. All questions were scaled from 1 to 5: (1 strongly agree; 2 agree; 3 neither agree nor disagree; 4 disagree; and 5 strongly disagree) .

ELIGIBILITY:
Inclusion Criteria:

* Children between (4-14 years) who underwent cochlear implantation surgery between 2015 and 2022.

Both sexes will be included.

Exclusion Criteria:

1. Patients with irregular device use.
2. Implantation less than 6 months.
3. Patients who refused to participate in the study.

Ages: 4 Years to 14 Years | Sex: All
Age Groups: Child
Study Population: Children between 4 to 14 years underwent cochlear implantation surgery between 2015 and 2022 in audiovestibular unit at Assiut University Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2023-03 (Estimated); Primary Completion 2023-05 (Estimated); Study Completion 2023-07 (Estimated)

PRIMARY OUTCOMES:
Parents' perspective Questionnaire | 2 years
  The outcome of CI surgery on Quality of Life (QoL) has been greatly investigated via parental questionnaire assessment. This questionnaire was designed with 11 subscales and 58 questions in total. All questions were scaled from 1 to 5: (1 strongly agree; 2 agree; 3 neither agree nor disagree; 4 disagree; and 5 strongly disagree)
Speech perception test with figures | 2 years

REFERENCES:
- [Background] Mulwafu W, Kuper H, Ensink RJ. Prevalence and causes of hearing impairment in Africa. Trop Med Int Health. 2016 Feb;21(2):158-65. doi: 10.1111/tmi.12640. Epub 2015 Dec 14. PMID 26584722
- [Background] Semaan MT, Fredman ET, Shah JR, Fares SA, Murray GS, Megerian CA. Surgical duration of cochlear implantation in an academic university-based practice. Am J Otolaryngol. 2013 Sep-Oct;34(5):382-7. doi: 10.1016/j.amjoto.2013.01.013. Epub 2013 Feb 13. PMID 23415572
- [Background] Niparko JK, Tobey EA, Thal DJ, Eisenberg LS, Wang NY, Quittner AL, Fink NE; CDaCI Investigative Team. Spoken language development in children following cochlear implantation. JAMA. 2010 Apr 21;303(15):1498-506. doi: 10.1001/jama.2010.451. PMID 20407059
- [Background] Ganek H, McConkey Robbins A, Niparko JK. Language outcomes after cochlear implantation. Otolaryngol Clin North Am. 2012 Feb;45(1):173-85. doi: 10.1016/j.otc.2011.08.024. Epub 2011 Oct 19. PMID 22115689
- [Background] Papsin BC, Gordon KA. Cochlear implants for children with severe-to-profound hearing loss. N Engl J Med. 2007 Dec 6;357(23):2380-7. doi: 10.1056/NEJMct0706268. No abstract available. PMID 18057340
- [Background] Hendriksma M, Bruijnzeel H, Bezdjian A, Kay-Rivest E, Daniel SJ, Topsakal V. Quality of life (QoL) evaluation of children using cochlear implants: agreement between pediatric and parent proxy-QoL reports. Cochlear Implants Int. 2020 Nov;21(6):338-343. doi: 10.1080/14670100.2020.1788858. Epub 2020 Jul 9. PMID 32643593
- [Background] Patrick DL, Edwards TC, Skalicky AM, Schick B, Topolski TD, Kushalnagar P, Leng M, O'Neill-Kemp AM, Sie KS. Validation of a quality-of-life measure for deaf or hard of hearing youth. Otolaryngol Head Neck Surg. 2011 Jul;145(1):137-45. doi: 10.1177/0194599810397604. PMID 21493349